CLINICAL TRIAL: NCT00158899
Title: A Multi-center, Three-staged With Interim Analyses, Parallel, Randomized, Double-blind, fenofibrate-and Placebo-controlled Proof of Concept and Dose-response Evaluation of the Safety, Tolerability, and Effects on Plasma High-density Lipoprotein Cholesterol (HDLc) and Triglycerides of Eight Weeks Treatment With GW501516 in Otherwise Healthy Patients With Low HDLc, Mildly to Moderately Elevated Triglycerides, and Normal Low-density Lipoprotein Cholesterol (LDLc)
Brief Title: GW501516 In Subjects Who Have Low Level Of High-Density Lipoprotein Cholesterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAD20001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Dyslipidaemias; Dyslipidaemia
Keywords: HDLc; high-density lipoprotein; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — GW 501516

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW501516 oral tablets

SUMMARY:
The purpose of this clinical research study is to compare up to 3 doses of an investigational drug GW501516 to placebo (an inactive pill that looks like GW501516) to see if it is safe, well tolerated and effective in improving (raising) low levels of "good cholesterol", high-density lipoprotein cholesterol (HDLc), as compared to placebo.

DETAILED DESCRIPTION:
A multicentre, two-staged with interim analysis, parallel, randomised, double blind, placebo-controlled, dose-ranging study of the safety, tolerability, and effects on plasma high-density lipoprotein cholesterol (HDLc) of 12 weeks treatment with 2.5mg, 5mg and 10mg daily doses of GW501516 in subjects with low HDLc

ELIGIBILITY:
Inclusion criteria:

* Have a fasting plasma HDLc concentration <=45mg/dL (<=1.16mmol/L), plasma LDLc levels that do not require treatment according to the National Cholesterol Education Program/Adult Treatment Panel III (NCEP/ATPÂ III) guidelines.
* Have a fasting plasma TG concentration =500mg/dL (=5.65mmol/L).

Exclusion criteria:

* Coronary heart disease.
* Diabetes mellitus.
* Atherosclerotic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2004-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The change from baseline in fasting plasma HDLc concentration at the end of 12 weeks of double-blind treatment. | 12 Weeks

SECONDARY OUTCOMES:
Changes from baseline at the end of 12 weeks of double-blind treatment of total cholesterol and other lipid parameters. Population pharmacokinetic parameters including oral clearance and apparent volume of distribution of GW501516. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MA, Study Director — GlaxoSmithKline
Locations (48):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- GSK Investigational Site, Hellerup, Denmark
- GSK Investigational Site, Tallinn, Estonia
- Finland (2):
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Tampere
- France (6):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Lagord
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Toulouse
- Germany (16):
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Koenigslutter, Lower Saxony
  - GSK Investigational Site, Winsen/Lohe, Lower Saxony
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Viersen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Netherlands (9):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Etten-Leur
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Rijswijk
  - GSK Investigational Site, Roelofarendsveen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Soerendonk
  - GSK Investigational Site, The Hague
- Norway (7):
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Soerumsand
  - GSK Investigational Site, Stavanger
- GSK Investigational Site, Coimbra, Portugal
- GSK Investigational Site, Malmo, Sweden